CLINICAL TRIAL: NCT01680263
Title: Kinesiotaping in Treatment of Pes Anserinus Tendino-bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kaynoosh Homayouni, Assistant professor of Physical Medicine and Rehabilitation, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K Homayouni
Record Dates: First submitted 2012-07-13; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Pes Anserinus Tendinobursitis
Keywords: Kinesiotaping; pes anserinus tendino-bursitis; nonsteroidal anti-inflammatory drugs; physical therapy
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesiotaping (Experimental): Use of kinesiotaping on the painful area in the form of "space correction". Kinesiotaping was repeated for 3 weeks with 1 week interval
  Interventions: Device: Kinesiotaping
- NSAIDs/Physical therapy (Active Comparator): treatment was done with NSAIDs and 10 sessions of daily physical therapy.
  Interventions: Procedure: NSAIDs/Physical therapy

INTERVENTIONS:
Device: Kinesiotaping — Use of kinesiotaping on the painful area in the form of "space correction". Kinesiotaping was repeated for 3 weeks with 1week interval
  Other Names: taping
  Arms: Kinesiotaping
Procedure: NSAIDs/Physical therapy — Use of non-steroidal anti-inflammatory drugs and 10 sessions of daily physical therapy.
  Other Names: non-steroidal anti-inflammatory drugs; physical therapy
  Arms: NSAIDs/Physical therapy

SUMMARY:
The aim of this study was to determine the effects of kinesiotaping in comparison to NSAIDs and physical therapy in treatment of pes anserinus tendino-bursitis.

DETAILED DESCRIPTION:
The treatment of pes anserinus tendino-bursitis includes refraining from aggravating activities, local modalities such as heat, ice, ultrasound (US), iontophoresis, phonophoresis, electrical stimulation (ES), nonsteroidal anti-inflammatory drugs (NSAIDs) and injections with either corticosteroids or local anesthetics. Another treatment that seems to have a significant effect on the improvement of the disease is kinesiotaping. Kinesiotaping is a cotton strip with an acrylic adhesive that is used for treating athletic injuries and a variety of physical conditions. The therapeutic effects of the tape is to relax the overused muscles and in rehabilitation to facilitate the underused muscles. Advocates claim that the wave pattern found on the kinesiotaping has a lifting effect on the skin which can diminish swelling and inflammation via improving circulation and reduce pain by removing pressure from pain receptors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of pes anserinus tendino-bursitis.

Exclusion Criteria:

* Previous history of trauma or surgery on the knee joint,
* History of NSAIDs induced acid-peptic disease
* Systemic and rheumatic diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pain (VAS)and swelling scores | 3 weeks
  Visual analog scale for pain evaluation Assessment of the local swelling via palpation

SECONDARY OUTCOMES:
The number of participants with adverse events | 3 weeks
  The number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kaynoosh Homayouni, M.D., Study Chair — Shiraz University of Medical Sciences; Shima Foruzi, M.D., Principal Investigator — Shiraz University of Medical Sciences; Fereshte Kalhori, M.D., Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Homayouni K, Foruzi S, Kalhori F. Effects of kinesiotaping versus non-steroidal anti-inflammatory drugs and physical therapy for treatment of pes anserinus tendino-bursitis: A randomized comparative clinical trial. Phys Sportsmed. 2016 Sep;44(3):252-6. doi: 10.1080/00913847.2016.1199251. Epub 2016 Jun 22. PMID 27276165